CLINICAL TRIAL: NCT01206803
Title: Polymorphisms of FSH Receptor, LH Receptor, LH and Ovarian Response to FSH in Controlled Ovarian Stimulation Using a GnRH Antagonist Protocol
Brief Title: Ovarian Response Prediction in In Vitro Fertilization (IVF) Patients
Status: Completed | Type: Observational
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Georg Griesinger, Prof. Dr. med. Georg Griesinger, M.Sc., University Hospital Schleswig-Holstein
Other Study IDs: GR 3422/3-1
Record Dates: First submitted 2010-09-21; First posted 2010-09-22 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Infertility, Subfertility
Keywords: ovarian stimulation; recombinant FSH; GnRH-antagonist; corifollitropin alfa
MeSH Terms: conditions — Infertility | interventions — Ovulation Induction; follitropin beta; ganirelix; Crinone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum samples for analysis of gonadotropins and Anti-Muellerian Hormone EDTA samples for DNA extraction
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Ovarian stimulation in a GnRH-antagonist protocol — Long-acting FSH 150µg & daily recombinant FSH 200 IU, GnRH-antagonist 0.25mg, 5,000-10,000 IU urinary hCG, triptorelin 0.2mg, vaginal progesterone
  Other Names: Elonva, Puregon, Orgalutran, Predalon, Crinone

SUMMARY:
The aim of the study is to explore ovarian response in terms of oocyte numbers after ovarian stimulation in a fixed gonadotropin dose GnRH-antagonist protocol by endocrine (AMH, FSH), demographic (age), sonographic (antral follicle count) and genetic factors (polymorphisms of gonadotropin receptors and secreted gonadotropins).

DETAILED DESCRIPTION:
Assisted reproduction by in-vitro fertilisation plays a pivotal role in the treatment of infertility, the understanding of reproductive biology, and future population dynamics. The success of assisted reproductive technologies (ART) is critically dependent on optimizing protocols for controlled ovarian stimulation which aim at providing an adequate number of good quality oocytes for in-vitro laboratory procedures. Interindividual variation in response to follicle-stimulating hormone (FSH) is a widespread problem with clinical and economical implications. A group of patients (9%-24%) tend to respond poorly to controlled ovarian stimulation (COS) whereas other patients tend to overrespond (2.5%) and thus run at risk of developing ovarian hyperstimulation syndrome, a potentially life-threatening disease. Polymorphisms of gonadotropin receptors seem to have an influence on the outcome of controlled ovarian hyperstimulation treatment, e.g. contributing to the variation in ovarian response to exogenous FSH between individuals. Other predictive factors include demographic (age), sonographic (follicular count in the ovaries, ovarian volume), endocrine (serum gonadotropin levels and Anti-Muellerian Hormone) and life-style factors (smoking, obesity). Such factors are routinely obtained prior to a treatment cycle, and are used to determine the optimal FSH starting dose or the best treatment regimen. The identification of gonadotropin receptor polymorphisms and variants in secreted gonadotropins prior to an ovarian stimulation treatment should allow the clinicians to tailor the starting dose of rFSH, especially for patients undergoing their first treatment cycle, as such ovarian response prediction will prevent cycle cancellations due to too low or too high ovarian response and reduce the risk of OHSS. The aim of the present study is to identify the prevalence of FSH and LH receptor polymorphisms and hormonal variants of LH and to study the variation attributable to these genetics factors when controlling for already established predictors of ovarian response to exogenous FSH in a multi-variate analysis.

ELIGIBILITY:
Inclusion Criteria:

Female patients for who the treating physician decides that treatment with long acting FSH 150µg in a GnRH-antagonist protocol is indicated.

Exclusion Criteria:

Contraindications for the use of gonadotropins (e.g., tumors, pregnancy/lactation, undiagnosed vaginal bleeding, hypersensitivity, ovarian cysts) Use of hormonal preparations within one month prior to inclusion

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Female patients with an indication for IVF or ICSI
Sampling Method: Probability Sample
Enrollment: 294 (Actual)
Dates: Start 2010-09; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
number of cumulus-oocyte-complexes | at the time of oocyte retrieval
  the number of 'oocytes' obtained by transvaginal retrieval after ovarian stimulation

CONTACTS AND LOCATIONS:
Locations (5):
- Germany (4):
  - Fertility Center Kiel, Kiel, S-H
  - University Hospital of Schleswig-Holstein, Campus Luebeck, Lübeck, Schleswig-Holstein
  - Prof. Axel Kamischke, Münster
  - Sabine Segerer, Würzburg
- Klinikk Hausken, Haugesund, Norway